CLINICAL TRIAL: NCT03942068
Title: Evaluating the Efficacy and Safety of Apatinib With Albumin-bound Paclitaxel in Patients With Platinum-resistant Recurrent Ovarian Cancer
Brief Title: Apatinib With Albumin-bound Paclitaxel in Patients With Platinum-resistant Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-HenanCH-OC019
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Albumin-Bound Paclitaxel; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- albumin-bound paclitaxel+apatinib (Experimental): albumin-bound paclitaxel:260mg/m2，q3w，d1 apatinib:500mg，qd，po
  Interventions: Drug: albumin-bound paclitaxel; Drug: Apatinib

INTERVENTIONS:
Drug: albumin-bound paclitaxel — Nanoparticle albumin-bound paclitaxel (nab-paclitaxel), a microtubule inhibitor
Drug: Apatinib — a novel oral antiangiogenic agent targeting vascular endothelial growth factor receptor (VEGFR2)

SUMMARY:
The study was designed to evaluate the efficacy and safety of apatinib with albumin-bound paclitaxel in patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
The study is an open, one-arm, prospec will collect 35 patients with platinum-resistant recurrent ovarian cancer treated with apatinib with albumin-bound paclitaxel from 2019 to 2020 in Henan Cancer Hospital.Antiangiogenic treatments have been implicated to play a major role in ovarian cancer (OC). Apatinib, a novel oral antiangiogenic agent targeting vascular endothelial growth factor receptor (VEGFR2), in combination with weekly paclitaxel, may improve clinical outcomes compared with apatinib or paclitaxel alone in patients with refractory or platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years and ≤70 years, signed informed consent.
2. Platinum resistant ovarian cancer (defined as relapsing within 6 months after the last administration of platinum-based chemotherapy) OR platinum refractory ovarian cancer (defined as progressing while on a platinum-based chemotherapy).
3. At least treated with one line of platinum-based chemotherapy.
4. Imaging confirmed diagnosis of progression occurred after the last treatment before enrollment.
5. Histologically or pathologically confirmed diagnosis of ovarian cancer as primary tumor.
6. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 version.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Patients must have a life expectancy of at least 3 months.
9. Patients must have adequate organ function as defined by the following criteria:
10. White blood cell count ≥ 3 x 10^9/L, Absolute neutrophil count (ANC) (≥ 1.5 x 10^9/L), Hemoglobin of ≥ 80 g/L, Platelets ≥ 70 x 10^9/L, Total bilirubin ≤ 1 x upper limit of normal (ULN), AST and ALT ≤ 2 x ULN, Serum creatinine ≤ 1 x ULN.

Exclusion Criteria:

* 1.Had prior exposure to apatinib or has known allegies to any of the excipients.

  2.Patients with trauma, surgical history, gastrointestinal bleeding, and melena within 1 month prior to treatment.

  3.Inadequately controlled hypertension. 4.History of abdominal fistula or gastrointestinal perforation within 28 days prior to Day 1.

  5.Imaging studies suggest that patients with tumors invading important blood vessels.

  6.Symptomatic central nervous system (CNS) metastasis. 7.History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months
  Objective Response Rate

SECONDARY OUTCOMES:
OS | through study completion, an average of 5 year
  Overall Survival
PFS | through study completion, an average of 5 year
  Progression-Free Survival
DCR | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months
  Disease Control Rate

IPD SHARING:
Plan to Share IPD: No